CLINICAL TRIAL: NCT04068623
Title: PERCEPTION Trial Protocol: Comparison of Predictive and Prognostic Capacities of Neutrophil, Lymphocyte and Platelet Counts and Tumour-infiltrating Lymphocytes in Triple Negative Breast Cancer
Brief Title: Correlation Between TILs and Blood Cell Counts in Triple Negative Breast Cancer Patients
Acronym: PERCEPTION
Status: Recruiting | Type: Observational
Sponsor: Centre Jean Perrin (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-A01861-56
Record Dates: First submitted 2019-07-31; First posted 2019-08-28 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Triple Negative Breast Cancer
Keywords: Triple negative breast cancer; NLR (Neutrophil-to-Lymphocyte Ratio); TILs (Tumor Infiltrating Lymphocytes); Peripheral blood cells
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma is collected in order to quantify the circulating tumor DNA at 1 year after the completion of radiation therapy and at the first metastatic recurrence
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Triple negative breast cancer
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Blood samples will be collected at 12 months after radiation therapy and at the time of first metastatic recurrence

SUMMARY:
The PERCEPTION study aims to assess the correlation between blood cell counts (Leucocytes, Neutrophils, Lymphocytes, Platelets, NLR (Neutrophil-to-Lymphocyte Ratio) and PLR (Platelet-to-Lymphocyte Ratio)) and Tumor Infiltrating Lymphocytes (TILs), at baseline and after surgery, for patients diagnosed with triple negative breast cancer. It also aims to assess these circulating elements and circulating tumor DNA as predictive factor of metastatic recurrence in triple negative breast cancer.

DETAILED DESCRIPTION:
Triple negative breast cancer (TNBC) is the most aggressive type of breast cancer. Because of the limited therapeutical strategies, early TNBC relapses are quite common during the five years following treatment.

It has been shown that the presence of tumor infiltrating lymphocytes (TILs) at baseline is related to good pathological response to neoadjuvant chemotherapy. In addition, the presence of a high quantity of TILs in the residual tumor after neoadjuvant chemotherapy is related to better survival rates.

Blood circulating elements, such as peripheral blood cells or circulating tumor DNA, could be of interest in predicting response to treatment and in the prediction of metastatic recurrences in different types of cancer, including breast cancer.

However, the correlation of these markers in triple negative breast cancer has not yet been thoroughly studied.

The PERCEPTION study aims to assess the correlation between blood cell counts (Leucocytes, Neutrophils, Lymphocytes, Platelets, NLR (Neutrophil-to-Lymphocyte Ratio) and PLR (Platelet-to-Lymphocyte Ratio)) and Tumor Infiltrating Lymphocytes (TILs), at baseline and after surgery, for patients diagnosed with triple negative breast cancer. It also aims to assess these circulating elements and circulating tumor DNA as predictive factor of metastatic recurrence in triple negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age > 18 years
* Diagnosed with primitive, non-metastatic, histologically proved, triple negative breast cancer
* Patient treated with chemotherapy, surgery and radiation therapy
* Patient able to understand the French language
* Patient affiliated to social security
* Obtaining signed written consent

Exclusion Criteria:

* Male
* Unavailable tumoral samples before inclusion
* Unavailable blood test results at baseline, before inclusion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women diagnosed and treated for non metastatic triple negative breast cancer
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2019-12-04 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2032-10 (Estimated)

PRIMARY OUTCOMES:
Assessment of the correlation between the lymphocyte infiltration rate assessed on biopsy, and the NLR (neutrophil-to-lymphocyte ratio) measured on blood samples, in women with triple negative breast cancer, at the time of diagnosis. | 3 years (the period of recruitment)
  * The value of NLR at diagnosis;
  * Tumor lymphocyte infiltration rate before treatment.

SECONDARY OUTCOMES:
Assessment of the correlation between the TILs assessed on biopsy, and the various parameters derived from the blood count (leucocytes, neutrophils, lymphocytes, platelets and PLR (Platelet-to-Lymphocyte Ratio)), at the time of diagnosis. | 3 years (the period of recruitment)
  * The values of leucocytes, lymphocytes, neutrophils, platelets and PLR at diagnosis;
  * Tumor lymphocyte infiltration rate before treatment
Assessment of the correlation between the various parameters derived from the blood count (leucocytes, neutrophils, lymphocytes, platelets, NLR and PLR) at the time of diagnosis, and the histological response to neo-adjuvant chemotherapy | 3 years (the period of recruitment)
  * The values of leucocytes, lymphocytes, neutrophils, platelets, NLR and PLR at diagnosis;
  * Histological response according to the Sataloff classification
Assessment of the correlation between the various parameters derived from the blood count (leucocytes, neutrophils, lymphocytes, platelets, NLR and PLR) at the time of diagnosis, and the TILs at surgery specimen after neoadjuvant chemotherapy. | 3 years (the period of recruitment)
  * The values of leucocytes, lymphocytes, neutrophils, platelets, NLR and PLR at diagnosis;
  * Tumor lymphocyte infiltration rate at surgery specimen
Assessment of the correlation between the various parameters derived from the blood count (leucocytes, neutrophils, lymphocytes, platelets, NLR and PLR) before surgery, and the lymphocyte infiltration rate at surgery after neoadjuvant chemotherapy. | 3 years
  * The values of leucocytes, lymphocytes, neutrophils, platelets, NLR and PLR before surgery;
  * Tumor lymphocyte infiltration rate at surgery specimen
Relationship between ctDNA and the metastatic relapse | 8 years
  * Measurement of plasma cDNA level
  * Metastatic relapse
Relationship between leucocyte value and the presence of circulating tumor DNA (ctDNA) | 8 years
  * The value of leucocytes
  * Measurement of plasma cDNA level
Relationship between lymphocyte value and the presence of circulating tumor DNA (ctDNA) | 8 years
  * The value of lymphocytes
  * Measurement of plasma cDNA level
Relationship between neutrophils value and the presence of circulating tumor DNA (ctDNA) | 8 years
  * The value of neutrophils
  * Measurement of plasma cDNA level
Relationship between platelet value and the presence of circulating tumor DNA (ctDNA) | 8 years
  * The value of platelets
  * Measurement of plasma cDNA level
Relationship between NLR value and the presence of circulating tumor DNA (ctDNA) | 8 years
  * The value of NLR
  * Measurement of plasma cDNA level
Relationship between PLR value and the presence of circulating tumor DNA (ctDNA) | 8 years
  * The value of PLR
  * Measurement of plasma cDNA level
Relationship between all the blood parameters and the metastatic relapse | 8 years
  * The values of leucocytes, lymphocytes, neutrophils, platelets, NLR and PLR
  * Metastatic relapse

CONTACTS AND LOCATIONS:
Overall Officials: Xavier DURANDO, Pr, Principal Investigator — Centre Jean Perrin
Locations (1):
- Centre Jean PERRIN, Clermont-Ferrand, Please Select, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lusho S, Durando X, Bidet Y, Molnar I, Kossai M, Bernadach M, Lacrampe N, Veyssiere H, Cavaille M, Gay-Bellile M, Radosevic-Robin N, Abrial C. PERCEPTION Trial protocol: Comparison of predictive and prognostic capacities of neutrophil, lymphocyte, and platelet counts and tumor-infiltrating lymphocytes in triple negative breast cancer. Medicine (Baltimore). 2020 Dec 11;99(50):e23418. doi: 10.1097/MD.0000000000023418. PMID 33327268